CLINICAL TRIAL: NCT02992509
Title: EMED Detruset Intravesical Electrical Stimulation Catheter for Treatment of Urge Urinary Incontinence and Overactive Bladder Syndrome in Females
Brief Title: IVES for Treatment of UUI and OAB
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Sam Siddighi, MD, Urogynecology/Pelvic Surgery, FPMRS, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5130321
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Urinary Bladder, Overactive; Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other): This pilot study group is a prospective observational study. It is not blinded and there is no control. This is a single arm study (treatment group) which will receive intravesical electrical stimulation with a total of 8 therapy sessions, each lasting 15 minutes. The sessions will be done in a serial fashion, 2 per week for 4 consecutive weeks.
  Interventions: Device: EMED detruset(TM) intravesical electrical stimulation

INTERVENTIONS:
Device: EMED detruset(TM) intravesical electrical stimulation — There will be a total of 8 therapy sessions, each lasting 15 minutes. The sessions will be done in a serial fashion, 2 per week for 4 consecutive weeks. The electrical parameters utilized will be those previously determined to be appropriate for OAB and UUI. As the beneficial effect of electrical stimulation is dependent on a "maximal" level of stimulation, the stimulation voltage will be increased during the first minute of treatment until the maximum tolerated by the patient is established and then backed-off by 1-2 Volts. The therapy will continue for 15 minutes in total for each session. The VAS will be marked by the patient before each treatment session throughout the therapy period, and other questionnaires will be administered.

SUMMARY:
The pilot study is intended to show the efficacy of intravesical electrical stimulation in treating overactive bladder with or without frequency and/or urgency urinary incontinence.

DETAILED DESCRIPTION:
The EMED Technologies detrusetTM intravesical electrical stimulation (IVES) catheter is indicated for use with the EMED detrusanTM 500 electrical generator for the treatment of overactive bladder and urge urinary incontinence (UI) in women who are not satisfied with or cannot tolerate other conservative treatments. EMED is interested in conducting a prospective randomized multi-center study of IVES therapy vs conventional UI treatments. In order to gain sufficient knowledge of the treatment effect and variability of IVES therapy to power an RCT, a pilot study will be initially conducted.

The pilot study is intended to show the efficacy of IVES in treating overactive bladder with or without frequency and/or urgency urinary incontinence with safety profile of IVES being no worse than with standard urological catheters.

A primary endpoint at 3 months showing reduction in incontinence events via a 7-level patient global impression of improvement will be established. Secondary endpoints will include PCI for subsets of symptoms, 3 day voiding diary, and patient satisfaction questionnaires.

Follow up at end of therapy and 3 months from the first therapy session will be conducted. 6-month, 9-month, and 12-month follow up can be conducted to establish durability of IVES therapy if it is found to be effective at 3 months after the first treatment

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-90 years old
* Urinary urge incontinence OR overactive bladder
* Prior trial of medical treatment for UUI or OAB

Exclusion Criteria:

* pelvic organ prolapse greater than stage 1
* multiple sclerosis
* parkinson's disease
* spinal cord injury
* long-term DM type I
* prior surgeries that may affect innervation of the detrusor nerves or the spinal cord
* pregnancy
* pacemaker/defibrillator
* PVR >150ml
* dementia
* Stress urinary incontinence
* intravesical botox injection within 1 year, PTNS within 6 months, or medical treatment for OAB within 3 weeks; bulking agent injection within 6 months

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reduction in incontinence | 3 months
  Primary endpoint is a reduction in incontinence events at 3 months post treatment as determined by a 7 point patient global impression of improvement

CONTACTS AND LOCATIONS:
Overall Officials: Sam Siddighi, MD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Background] Hagerty JA, Richards I, Kaplan WE. Intravesical electrotherapy for neurogenic bladder dysfunction: a 22-year experience. J Urol. 2007 Oct;178(4 Pt 2):1680-3; discussion 1683. doi: 10.1016/j.juro.2007.03.188. Epub 2007 Aug 17. PMID 17707024
- [Background] Cheng EY, Richards I, Balcom A, Steinhardt G, Diamond M, Rich M, Donovan JM, Carr MC, Reinberg Y, Hurt G, Chandra M, Bauer SB, Kaplan WE. Bladder stimulation therapy improves bladder compliance: results from a multi-institutional trial. J Urol. 1996 Aug;156(2 Pt 2):761-4. PMID 8683778
- [Background] Hong CH, Lee HY, Jin MH, Noh JY, Lee BH, Han SW. The effect of intravesical electrical stimulation on bladder function and synaptic neurotransmission in the rat spinal cord after spinal cord injury. BJU Int. 2009 Apr;103(8):1136-41. doi: 10.1111/j.1464-410X.2008.08189.x. Epub 2008 Nov 18. PMID 19021629
- [Background] Lombardi G, Musco S, Celso M, Ierardi A, Nelli F, Del Corso F, Del Popolo G. Intravesical electrostimulation versus sacral neuromodulation for incomplete spinal cord patients suffering from neurogenic non-obstructive urinary retention. Spinal Cord. 2013 Jul;51(7):571-8. doi: 10.1038/sc.2013.37. Epub 2013 Apr 30. PMID 23628893